CLINICAL TRIAL: NCT02011880
Title: Standardization Research of TCM Syndrome Differentiation and Treatment on Advanced Breast Cancer
Status: Temporarily not available | Type: Expanded Access
Sponsor: Shanghai University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: ZYSNXD-CC-ZDYJ043
Record Dates: First submitted 2013-12-10; First posted 2013-12-13 (Estimated); Last update posted 2013-12-13 (Estimated); Status verified 2013-09

CONDITIONS: Breast Cancer; Bone Metastasis
Keywords: breast cancer; bone metastasis; traditional Chinese medicine(TCM)
MeSH Terms: conditions — Breast Neoplasms

INTERVENTIONS:
Dietary Supplement: Chinese Herbs — Dietary Supplement:Experiment group:
  Fructus Cnidii,Psoralea Corylifolin L.，monkshood
  -Granules,Oral(add into the breast cancer postoperative prescription solution),A Pack(Fructus Cnidii 9g，Psoralea Corylifolin L. 15g，monkshood 9g),Bid Days,3 Periods(a month is a period),Until progression/unacceptable toxicity
  Breast Cancer Postoperative Prescription
  -Water Decoction,Oral,200ml,Bid Days,3 Periods(a month is a period),Until progression/unacceptable toxicity
  Dietary Supplement:Contrast Group:
  Breast Cancer Postoperative Prescription
  -Water Decoction,Oral,200ml,Bid Days,3 Periods( a month is a period),Until progression/unacceptable toxicity
  Other Names: Fructus Cnidii; Psoralea Corylifolin L.; monkhsood; Breast Cancer Postoperative Prescription

SUMMARY:
The purpose of this clinical research study is to learn if the clinical effects of combined Chinese herbal medicine with endocrine therapy is better than endocrine therapy alone in improving the quality of life and shrinking and slowing the growth of the cancer in women with breast cancer bone metastasis.

DETAILED DESCRIPTION:
OBJECTIVES:

* Evaluate the effect of the Chinese herbal medicine on relieving the bone pain for patients with breast cancer bone metastasis.
* Evaluate the effect of the Chinese herbal medicine on improving the quality of life and shrinking and slowing the growth of the cancer in women with breast cancer bone metastasis.

OUTLINE: This is a randomized,multicentric, placebo-controlled, double-blind study. Patients are dynamic randomized to one of two treatment arms.

* Arm I:Patients receive traditional Chinese medicine(trial drugs) and endocrine therapy for 3 months.
* Arm II:Patients receive placebo and endocrine therapy for 3 months. All patients will be followed up for another 3 months with the trial drugs and endocrine therapy.

According to the sample size estimate:There are 296 patients (148 per treatment arm)will be collected in this trial.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed breast cancer and hormone receptor positive.
* Bone metastasis and have a measurable foci.
* TCM syndrome type is deficiency of both vital energy and Yin ;maladjustment of ChongRen with deficiency Yang syndrome.
* The Karnofsky score ≥60.
* VAS score ≥3.
* Expected survival at least 6 months or greater.
* Age between 20 to 70(include 20 and 70).
* The function of cardiovascular,hepar,renal and hematopoieses is relatively normal.

Exclusion Criteria:

* Women during the pregnancy or breast feeding.
* With a cardiovascular,hepar,renal,hematopoieses or other serious complications.
* Be allergic to the trial drugs.
* Participating in other trials.

Ages: 20 Years to 70 Years | Sex: Female
Age Groups: Adult, Older Adult